CLINICAL TRIAL: NCT02941588
Title: The Impact of Early Surgery and Maintenance of Antiplatelet Therapy on Intraoperative Bleeding and Major Adverse Cardiovascular Event After Percutaneous Coronary Intervention
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Won Ho Kim, MD, Clinical Associate Professor, Seoul National University Hospital
Other Study IDs: 1604-023-753
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Acute Coronary Syndrome; Drug-eluting Stent; Aspirin
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- non-cardiac surgery after DES: The patients who underwent non-cardiac surgery after percutaneous coronary intervention with drug-eluting stent
  Interventions: Procedure: Non-cardiac surgery

INTERVENTIONS:
Procedure: Non-cardiac surgery — Any surgery with general anesthesia except cardiac surgery

SUMMARY:
Recent guidelines of the ACC/AHA suggest that elective non-cardiac surgery (NCS) should optimally be delayed one year after percutaneous coronary intervention (PCI) with drug-eluting stent (DES). Regarding the antiplatelet agents, dual antiplatelet therapy, or at least aspirin is recommended to be continued considering the relative risk of bleeding and stent thrombosis especially during the first 4 to 6 weeks after DES implantation. However, these recommendations are based upon insufficient and conflicting evidences.

DETAILED DESCRIPTION:
Recent guidelines of the ACC/AHA suggest that elective non-cardiac surgery (NCS) should optimally be delayed one year after percutaneous coronary intervention (PCI) with drug-eluting stent (DES). Regarding the antiplatelet agents, dual antiplatelet therapy, or at least aspirin is recommended to be continued considering the relative risk of bleeding and stent thrombosis especially during the first 4 to 6 weeks after DES implantation. However, these recommendations are based upon insufficient and conflicting evidences.

The aim of our study was (1) to determine independent risk factors for postoperative adverse events and the strength of their association, (2) to assess the incidences of postoperative morbidities including major adverse cardiovascular and cerebral event as a function of time between PCI and surgery and (3) to compare bleeding amount and transfusion requirements between different intervals from PCI to surgery and durations of antiplatelet agent administration prior to surgery. To achieve this aim, we undertook a retrospective cohort study of the patients who underwent noncardiac surgery after PCI with DES.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent non-cardiac surgery within 5 years after percutaneous coronary intervention with drug-eluting stent at Seoul National University Hospital between April 2004 and August 2017

Exclusion Criteria:

* Patients who underwent percutaneous coronary intervention with balloon angioplasty or bare metal stent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent non-cardiac surgery within 5 years after percutaneous coronary intervention with drug-eluting stent at Seoul National University Hospital between April 2004 and August 2017
Sampling Method: Non-Probability Sample
Enrollment: 1582 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebral event | during postoperative 30 days
  a composite of non-fatal myocardial infarction, coronary revascularization, pulmonary embolism and stroke

SECONDARY OUTCOMES:
Composite morbidity | during postoperative 30 days
  composite of overall postoperative morbidity, including Major adverse cardiovascular and cerebral event and all respiratory, cardiac, renal and other complications during postoperative 30 days.
Major bleeding event | during the 24 hours from the surgery
  a bleeding event with any one of the following (1) A preoperative hematocrit ≤ 30% or a drop of hematocrit ≥10% as well as transfusion of ≥2 units of RBC during the surgery, or (2) the patient received a transfusion of ≥4 units of red blood cells within a 24 hour period, or (3) any one of the following interventions (i.e., embolization, superficial vascular repair, nasal packing); or retroperitoneal, intraspinal or intraocular bleeding (confirmed clinically or on imaging).

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No